CLINICAL TRIAL: NCT05088148
Title: Comparison of Pesticide and Pharmaceutical Contaminants Levels in Placenta and Cord Blood Samples of Pregnant Women With Fetal Growth Retardation and Healthy Pregnant Women
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Sponsor
Other Study IDs: Kutahya Health Sciences Uni
Record Dates: First submitted 2021-10-11; First posted 2021-10-21 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2021-10

CONDITIONS: Fetal Growth Retardation
MeSH Terms: conditions — Fetal Growth Retardation | interventions — Pesticides

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — placenta and cord blood samples of pregnant women
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: FGR group: Estimated fetal weight <10th percentile
  Interventions: Other: . Pesticide and Pharmaceutical analysis
- Group 2: Control group: Healthy pregnants who will give birth 37th and after gestational week
  Interventions: Other: . Pesticide and Pharmaceutical analysis

INTERVENTIONS:
Other: . Pesticide and Pharmaceutical analysis — Pesticide and Pharmaceutical analysis will be done with LC-MS/MS device.

SUMMARY:
Aim: In this study, pesticide and pharmaceutical contaminants levels in the placenta and cord blood of pregnant women with fetal growth retardation and healthy pregnant women will be compared in placenta and cord blood samples after delivery.

DETAILED DESCRIPTION:
The study will be conducted with a total of 40 pregnant women, 20 of whom are in the control groups and those with FGR diagnoses. Cases in both groups will be matched in terms of demographic information. Demographic information (including socioeconomic status, educational level, region of residence), ultrasound and Doppler examination results, newborn weight at birth, APGAR score, gender, mode of delivery, whether there is a need for neonatal intensive care or not will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-40 years
* Gestational age between 320/7 - 396/7 weeks
* Singleton pregnancy
* For the FGR group: estimated fetal weight <10th percentile
* For the control group: being healthy pregnant
* Intact amniotic membrane

Exclusion Criteria:

* Multiple pregnancies
* Cardiovascular disease
* Chronic hypertension
* Autoimmune disease
* Intrahepatic cholestasis of pregnancy
* Preeclampsia-eclampsia
* Sepsis
* Placenta accreta spectrum
* Abnormalities of placenta
* The chromosomal or congenital structural anomaly of the fetus
* Smoking
* BMI >30 kg/m2

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant
Study Population: The study will be conducted with a total of 40 pregnant women, 20 of whom are in the control groups and those with FGR diagnoses. Cases in both groups will be matched in terms of demographic information. Demographic information (including socioeconomic status, educational level, region of residence), ultrasound and Doppler examination results, newborn weight at birth, APGAR score, gender, mode of delivery, whether there is a need for neonatal intensive care or not will be recorded.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-03-29 (Estimated); Primary Completion 2023-02-26 (Estimated); Study Completion 2023-03-26 (Estimated)

PRIMARY OUTCOMES:
Pesticide and Pharmaceutical analysis | 1 year
  Pesticide and pharmaceutical contaminants levels in pregnant women's placenta and cord blood will be measured in placenta and cord blood samples after delivery.

SECONDARY OUTCOMES:
Multi logistic regression analysis. | 1 month
  If there is a significant difference in other data, including the pesticide and pharmaceutical contaminants levels, in the FGR group, the effect of each factor on the development of FGR will be analyzed by multi logistic regression analysis.
ROC analysis | 1 month
  If the pesticide and pharmaceutical contaminants levels is found to be significantly higher in the FGR group, the cut-off value will be obtained by ROC analysis.